CLINICAL TRIAL: NCT06853964
Title: A Study to Evaluate the Safety and Effectiveness of AlloMend® Acellular Dermal Matrix Used in Post Mastectomy Pre-Pectoral Breast Reconstruction and Followed for Up To 12-Months Post-Operatively
Brief Title: Retrospective Study of AlloMend Acellular Dermal Matrix (ADM) Allograft and Pre-Pectoral Breast Reconstruction
Status: Active, not recruiting | Type: Observational
Sponsor: AlloSource (Industry)
Responsible Party: Sponsor
Other Study IDs: ADM2024-001
Record Dates: First submitted 2024-11-19; First posted 2025-03-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pre-Pectoral Breast Reconstruction Following Mastectomy
Keywords: AlloMend; Acellular Dermal Matrix; Pre-pectoral Breast Reconstruction; Allografts

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: AlloMend® Acellular Dermal Matrix allograft — AlloSource, a non-profit supplier of allografts and one of the nation's leading tissue banks, introduced AlloMend® Acellular Dermal Matrix allograft to bring the benefits of regenerative medicine to more patients. cellular allograft matrices, unlike synthetic materials or xenografts, are recognized as human tissue by the body for graft incorporation by the recipient, minimizing the risk of inflammation or rejection. AlloMend® Acellular Dermal Matrix allograft has been shown to incorporate into the surgical site and demonstrates blood vessel infiltration.

SUMMARY:
This retrospective, single-site study will provide information regarding the efficiency of AlloMend® Acellular Dermal Matrix allograft in Pre-Pectoral Breast Reconstruction surgery following a single or double mastectomy.

DETAILED DESCRIPTION:
AlloMend® Acellular Dermal Matrix AlloMend® is a sterile, ready-to-use, human-derived acellular dermal matrix (ADM) allograft that can be used in a number of reconstructive and other surgical procedures. It is made from donated human full-thickness skin. After the epidermal and hypodermal layers are removed, the tissue is treated by a proprietary cleansing process.

AlloMend® is intended to be used in conjunction with a breast implant or tissue expander to stabilize implant position and minimize implant loss during post-single or double mastectomy, unilateral or bilateral pre-pectoral breast reconstruction in women 18 years of age or older. AlloMend® may be used in either one-stage (direct-to-implant) or two-stage (expander-to-implant) procedures.

This retrospective study will be performed at one center in the United States.

Information from the preoperative clinical visit and Pre-Pectoral Breast Reconstruction surgery utilizing AlloMend® Acellular Dermal Matrix allograft, approximately 200 breasts (and up to 100 patients), and the follow-up clinical visits at approximately 2 weeks, 6 weeks, 3 months, 6 months, and 12 months, including clinical assessments, imaging, and patient-reported outcomes, will be collected.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following inclusion criteria to participate in this study:

* Female ≥ 18 years old.
* Patients have undergone a single or double mastectomy, followed by AlloMend® Acellular Dermal Matrix -assisted, pre-pectoral breast reconstruction.
* Patients have undergone either one-stage (direct-to-implant) or two-stage (expander-to-implant), unilateral or bilateral pre-pectoral breast reconstruction using AlloMend®.

Exclusion Criteria:

Patients must not meet any of the following criteria to be considered for this clinical trial:

* Did not utilize AlloMend® Acellular Dermal Matrix allograft during pre-pectoral breast reconstruction
* Did not have post-operative evaluations at the clinical site.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who require a single or double mastectomy and have undergone Pre-Pectoral Breast Reconstruction surgery with the use of AlloMend® Acellular Dermal Matrix allograft are eligible to participate. Patients who meet all the inclusion criteria but do not meet any of the exclusion criteria are eligible to enter the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective Analysis of Clinical and Surgical Outcomes in Pre-Pectoral Breast Reconstruction with AlloMend® | Up to 12-month post-operatively
  This primary outcome measure will retrospectively collect descriptive data on patients who have undergone single or double mastectomy followed by pre-pectoral breast reconstruction using AlloMend® Acellular Dermal Matrix allograft. Data will be extracted from medical records and will include patient demographics, medical history, surgical techniques, intraoperative and postoperative complications, prescribed medications, and adjuvant treatments such as chemotherapy and radiation. The objective is to characterize patient profiles, surgical outcomes, and potential complications associated with this reconstructive approach.

SECONDARY OUTCOMES:
Retrospective Evaluation of Follow-Up Clinical, Imaging, and Surgical Outcomes | Up to 12-month post-operatively
  This outcome measure will retrospectively assess post-treatment follow-up data, including physical examinations, imaging findings, physical therapy progress, and the incidence of revision surgery. Data will be extracted from patient records to evaluate recovery progress, functional improvements, and any complications or need for additional interventions.
Retrospective Assessment of Patient-Reported Health Status and Quality of Life | Up to 12 months
  This outcome measure will retrospectively evaluate patients' self-reported overall health status and quality of life following surgical intervention. Data will be collected from existing medical records, including patient-reported responses and clinical interviews, to assess perceived well-being, functional limitations, pain levels, and overall satisfaction with treatment outcomes. No specific tool was used to gather their responses.

CONTACTS AND LOCATIONS:
Locations (1):
- Janiga MDs Plastic Surgery and Cosmetic Center, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No